CLINICAL TRIAL: NCT03861936
Title: BOTOX® (onabotulinumtoxinA) Treatment of Masseter Muscle Prominence: A Phase 2b, Multicenter, Randomized, Double-Blind, Multi-Dose, Placebo-Controlled Study
Brief Title: BOTOX® (onabotulinumtoxinA) Treatment of Masseter Muscle Prominence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1789-202-008
Record Dates: First submitted 2019-02-25; First posted 2019-03-05 (Actual); Results first posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Masseter Muscle Prominence
MeSH Terms: interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BOTOX® 72U (Experimental): OnabotulinumtoxinA (botulinum toxin Type A; BOTOX®) 72 units (U) total dose administered intramuscularly to the bilateral masseter muscles on Day 1.
  Interventions: Biological: OnabotulinumtoxinA
- BOTOX® 48U (Experimental): OnabotulinumtoxinA (botulinum toxin Type A; BOTOX®) 48U total dose administered intramuscularly to the bilateral masseter muscles on Day 1.
  Interventions: Biological: OnabotulinumtoxinA
- Placebo (Placebo Comparator): Placebo (Normal saline) administered intramuscularly to the bilateral masseter muscles on Day 1.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Biological: OnabotulinumtoxinA — OnabotulinumtoxinA (botulinum toxin Type A;BOTOX®) administered intramuscularly to the bilateral masseter muscles on Day 1.
  Other Names: BOTOX®; botulinum toxin Type A
  Arms: BOTOX® 48U; BOTOX® 72U
Drug: Normal saline — Normal saline (placebo) administered intramuscularly to the bilateral masseter muscles on Day 1.
  Arms: Placebo

SUMMARY:
Based on the results of the Phase 2 Study 191622-130 [NCT02010775], the current Phase 2b study is designed to further evaluate the safety and efficacy of BOTOX® for the treatment of Masseter Muscle Prominence (MMP) in adults.

ELIGIBILITY:
Inclusion Criteria

* Participant has bilateral MMP (identical grades for left and right masseter), as determined at the Day 1 visit by the investigator using the MMPS
* Participant has bilateral MMP, as determined at the Day 1 visit by the participant using the Masseter Muscle Prominence Scale-Participant (MMPS-P)
* Body mass index (BMI) ≤ 30 kilogram/square meter (kg/m^2) using the calculation: BMI = weight (kg) [height (m^2)]
* Female participants willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up period. A female participant is eligible to participate if she is not pregnant (has a negative urine pregnancy result prior to randomization), not breastfeeding, and at least one of the following conditions applies:

  1. Not a woman of childbearing potential (WOCBP) OR
  2. A WOCBP who agrees to follow the contraceptive guidance during the treatment and follow-up period
* Able, as assessed by the investigator, and willing to follow study instructions and likely to complete all required study visits.

Exclusion Criteria

* Any medical condition that may put the participant at increased medical risk with exposure to BOTOX®, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function
* Any uncontrolled medical condition
* An anticipated need for surgery or overnight hospitalization during the study
* An anticipated need for treatment with botulinum toxin of any serotype for any indication during the study (other than study intervention)
* History of dental or surgical procedure for lower facial shaping or masseter muscle reduction
* Prior mid-facial and/or lower facial treatment with nonpermanent soft tissue fillers, synthetic implantations, autologous fat transplantation, fat-reducing injectables, and/or skin-tightening laser treatments within 6 months of entry into the study
* Current or planned dental or facial procedures during the study period (eg, braces, dental implants, and reconstructive or aesthetic surgery) that could interfere with MMPS, as determined by the investigator
* Facial hair or scarring (eg, acne) significant enough to interfere with the 3D clinical photography assessment
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study
* Prior exposure to botulinum toxin of any serotype to the masseter muscle or lower face at any time, or to any other part of the body within the 6 months prior to Day 1
* Current intraoral infection, including infection of the mouth or gums, or facial skin infection requiring medical treatment in the opinion of the investigator
* History of or current Temporomandibular Joint Dysfunction (TMJD), or presence of signs/symptoms of possible TMJD, in the opinion of the investigator
* Weakness of the masseter, pterygoid, or temporalis muscles due to trauma, facial nerve injury, or other condition that could interfere with normal chewing and jaw clenching, as determined by the investigator
* Excess lower facial fat, loose or lax skin in lower face, or parotid gland prominence that could interfere with MMPS, as determined by the investigator
* Significant asymmetry of left and right sides of the face that could prevent identical MMPS grading on both sides of the face, as determined by the investigator
* Masseter prominence due to other etiologies (eg, parotid gland infection, parotiditis, malignancy) based upon findings from the oral examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Brandstetter, Study Director — Allergan
Locations (14):
- United States (14):
  - Total Skin & Beauty Dermatology Center, PC, Birmingham, Alabama
  - Westside Aesthetics, Los Angeles, California
  - Skin Care and Laser Physicians of Beverly Hills, Los Angeles, California
  - Cosmetic Laser Dermatology, San Diego, California
  - Baumann Cosmetic and Research Institute, Miami, Florida
  - DeNova Research, Chicago, Illinois
  - Etre, Cosmetic Dermatology and Laser Center, New Orleans, Louisiana
  - Saint Louis University Dermatology, St Louis, Missouri
  - Skin Specialists, PC, Omaha, Nebraska
  - Nashville Centre for Laser and Facial Surgery, Nashville, Tennessee
  - DermResearch, Inc., Austin, Texas
  - Bellaire Dermatology Associates, Bellaire, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - Advanced Clinical Research Gateway Aesthetic Institute & Laser Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Allergan will share de-identified patient-level data and study-level data including protocols and clinical study reports for phase 2 - 4 trials completed after 2008 that are registered to ClinicalTrials.gov or EudraCT, have received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published. To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes. More information can be found on http://www.allerganclinicaltrials.com/.
Supporting Information: Study Protocol, CSR
Time Frame: After having received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published.
Access Criteria: To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes.
URL: http://www.allerganclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- BOTOX® 48U: OnabotulinumtoxinA (botulinum toxin Type A; BOTOX®) 48 units (U) total dose administered intramuscularly to the bilateral masseter muscles on Day 1.
- BOTOX® 72U: OnabotulinumtoxinA (botulinum toxin Type A; BOTOX®) 72U total dose administered intramuscularly to the bilateral masseter muscles on Day 1.
Period: Overall Study
Arm/Group | Placebo | BOTOX® 48U | BOTOX® 72U
Started | 48 | 53 | 49
Completed | 34 | 43 | 39
Not Completed | 14 | 10 | 10
Not completed — Withdrawal by Subject | 4 | 1 | 3
Not completed — Lost to Follow-up | 5 | 3 | 3
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Protocol Deviation | 0 | 0 | 1
Not completed — Reason not Specified | 5 | 5 | 3

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-treat (mITT) Population consisted of all randomized participants who received study treatment and had at least 1 postbaseline Masseter Muscle Prominence Scale (MMPS) assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BOTOX® 48U | BOTOX® 72U | Total
Number analyzed (Participants) | 46 | 53 | 46 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (12.11) | 38.3 (10.50) | 38.9 (10.60) | 39.3 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 45 | 42 | 130
  Male | 3 | 8 | 4 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 13 | 9 | 26
  Not Hispanic or Latino | 42 | 40 | 37 | 119
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 7 | 8 | 10 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Black or African American | 2 | 1 | 3 | 6
  White | 36 | 42 | 32 | 110
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Masseter Muscle Prominence Scale (MMPS) Grade ≤ 3 at Day 90 as Assessed by the Investigator
Description: The investigator assessed the severity of the participant's masseter muscle prominence (MMP) using the MMPS 5-point scale where: 1=minimal (best), 2=mild, 3=moderate, 4=marked, and 5=very marked (worst). The percentage of participants where the investigator selected 1=minimal, 2=mild, or 3=moderate are reported.
Time Frame: Day 90
Population: mITT Population consisted of all randomized participants who received study treatment and had at least 1 postbaseline MMPS assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX® 48U | BOTOX® 72U
Number analyzed (Participants) | 46 | 53 | 46
percentage of participants | 21.7 [9.8 to 33.7] | 90.6 [82.7 to 98.4] | 91.3 [83.2 to 99.4]
Statistical Analysis 1: Comparison: Placebo vs BOTOX® 48U; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel — P-values for between-treatment comparisons are based on Cochran-Mantel-Haenszel (CMH) model stratified by baseline MMPS Grade (4 or 5); Percentage Difference = 68.8, 95% CI 2-sided [54.5 to 83.1]
Statistical Analysis 2: Comparison: Placebo vs BOTOX® 72U; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel — P-values for between-treatment comparisons are based on CMH model stratified by baseline MMPS Grade (4 or 5); Percentage Difference = 69.6, 95% CI 2-sided [55.1 to 84.0]

2. Primary Outcome: Number of Participants With at Least One Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. A TEAE is an AE that occurs or worsens after receiving study drug.
Time Frame: First dose (Day 1) to the End of Study (Up to Day 180)
Population: Safety Population consisted of all participants who received at least 1 injection of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BOTOX® 48U | BOTOX® 72U
Number analyzed (Participants) | 48 | 53 | 49
Participants | 12 | 18 | 14

3. Primary Outcome: Change From Baseline in Systolic Blood Pressure
Time Frame: Baseline (Day 1) to the End of Study (Up to Day 180)
Population: Safety Population consisted of all participants who received at least 1 injection of study intervention. Number analyzed is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | BOTOX® 48U | BOTOX® 72U
Number analyzed (Participants) | 48 | 53 | 49
millimeters of mercury (mmHg)
  Baseline | 115.8 (13.52) | 118.6 (10.39) | 114.7 (13.64)
  Change from Baseline to End of Study: number analyzed (Participants) | 47 | 53 | 48
  Change from Baseline to End of Study | -0.3 (10.09) | -1.2 (12.05) | -0.3 (10.82)

4. Primary Outcome: Change From Baseline in Diastolic Blood Pressure
Time Frame: Baseline (Day 1) to the End of Study (Up to Day 180)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | BOTOX® 48U | BOTOX® 72U
Number analyzed (Participants) | 48 | 53 | 49
mmHg
  Baseline | 76.8 (8.28) | 77.7 (8.63) | 76.6 (10.09)
  Change from Baseline to End of Study: number analyzed (Participants) | 47 | 53 | 48
  Change from Baseline to End of Study | 0.1 (6.72) | -0.2 (8.07) | 0.8 (9.44)

5. Primary Outcome: Change From Baseline in Respiratory Rate
Description: Respiratory rate is calculated as number of breaths (inhalation and exhalation) in one minute.
Time Frame: Baseline (Day 1) to the End of Study (Up to Day 180)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | Placebo | BOTOX® 48U | BOTOX® 72U
Number analyzed (Participants) | 48 | 53 | 49
breaths/minute
  Baseline | 15.5 (2.01) | 15.6 (2.14) | 15.2 (1.92)
  Change from Baseline to End of Study: number analyzed (Participants) | 47 | 53 | 48
  Change from Baseline to End of Study | 0.1 (1.75) | 0.1 (1.85) | 0.1 (1.66)

6. Primary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate measures the number of times your heart beats per minute.
Time Frame: Baseline (Day 1) to the End of Study (Up to Day 180) ]
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Placebo | BOTOX® 48U | BOTOX® 72U
Number analyzed (Participants) | 48 | 53 | 49
beats/minute
  Baseline | 76.9 (12.47) | 73.9 (10.83) | 74.2 (11.22)
  Change from Baseline to End of Study: number analyzed (Participants) | 47 | 53 | 48
  Change from Baseline to End of Study | -0.2 (10.69) | -0.8 (9.83) | 0.9 (10.59)

7. Secondary Outcome: Percentage of Participants Who Achieved Participant Masseter Muscle Prominence Scale-Participant (MMPS-P) Grade ≤ 3 at Day 90 as Assessed by the Participant
Description: The participant assessed the severity of their MMP using the MMPS-P 5-point scale where: 1=not at all pronounced (best), 2=mildly pronounced, 3=moderately pronounced, 4=pronounced, and 5=very pronounced (worst). The percentage of participants who selected 1=not at all pronounced, 2=mildly pronounced, or 3=moderately pronounced are reported.
Time Frame: Day 90
Population: mITT Population consisted of all randomized participants who received study treatment and had at least 1 postbaseline MMPS assessment. Missing postbaseline data are imputed using last observation carried forward (LOCF).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX® 48U | BOTOX® 72U
Number analyzed (Participants) | 46 | 53 | 46
percentage of participants | 47.8 [33.4 to 62.3] | 96.2 [91.1 to 100.0] | 93.5 [86.3 to 100.0]
Statistical Analysis 1: Comparison: Placebo vs BOTOX® 48U; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel — P-values for between-treatment comparisons are based on CMH model stratified by baseline MMPS Grade (4 or 5); Percentage Difference = 48.4, 95% CI 2-sided [33.1 to 63.7]
Statistical Analysis 2: Comparison: Placebo vs BOTOX® 72U; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel — P-values for between-treatment comparisons are based on CMH model stratified by baseline MMPS Grade (4 or 5); Percentage Difference = 45.7, 95% CI 2-sided [29.5 to 61.8]

8. Secondary Outcome: Percentage of Participants Who Achieved ≥ 2-grade MMPS Improvement From Baseline at Day 90 as Assessed by the Investigator
Description: The investigator assessed the severity of the participant's MMP using the MMPS 5-point scale where: 1=minimal (best), 2=mild, 3=moderate, 4=marked, and 5=very marked (worst). The percentage of participants who achieved a ≥ 2-grade improvement (decrease) from Baseline as assessed by the investigator are reported.
Time Frame: Baseline (Day 1) to Day 90
Population: mITT Population consisted of all randomized participants who received study treatment and had at least 1 postbaseline MMPS assessment. Missing postbaseline data are imputed using LOCF.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX® 48U | BOTOX® 72U
Number analyzed (Participants) | 46 | 53 | 46
percentage of participants | 10.9 [1.9 to 19.9] | 66.0 [53.3 to 78.8] | 71.7 [58.7 to 84.8]
Statistical Analysis 1: Comparison: Placebo vs BOTOX® 48U; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel — P-values for between-treatment comparisons are based on CMH model stratified by baseline MMPS Grade (4 or 5); Percentage Difference = 55.2, 95% CI 2-sided [39.6 to 70.8]
Statistical Analysis 2: Comparison: Placebo vs BOTOX® 72U; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel — P-values for between-treatment comparisons are based on CMH model stratified by baseline MMPS Grade (4 or 5); Percentage Difference = 60.9, 95% CI 2-sided [45.1 to 76.7]

9. Secondary Outcome: Percentage of Participants Who Achieved ≥ 2-grade MMPS-P Improvement From Baseline at Day 90 as Assessed by the Participant
Description: The participant assessed the severity of their MMP using the MMPS-P 5-point scale where: 1=not at all pronounced (best), 2=mildly pronounced, 3=moderately pronounced, 4=pronounced, and 5=very pronounced (worst). The percentage of participants who achieved a ≥ 2-grade improvement (decrease) from Baseline as assessed by the participant are reported.
Time Frame: Baseline (Day 1) to Day 90
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX® 48U | BOTOX® 72U
Number analyzed (Participants) | 46 | 53 | 46
percentage of participants | 32.6 [19.1 to 46.2] | 86.8 [77.7 to 95.9] | 80.4 [69.0 to 91.9]
Statistical Analysis 1: Comparison: Placebo vs BOTOX® 48U; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel — P-values for between-treatment comparisons are based on CMH model stratified by baseline MMPS Grade (4 or 5); Percentage Difference = 54.2, 95% CI 2-sided [37.9 to 70.5]
Statistical Analysis 2: Comparison: Placebo vs BOTOX® 72U; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel — P-values for between-treatment comparisons are based on CMH model stratified by baseline MMPS Grade (4 or 5); Percentage Difference = 47.8, 95% CI 2-sided [30.1 to 65.6]

10. Secondary Outcome: Percentage of Participants Who Achieved Participant Self-Assessment of Change (PSAC) in MMP Grade ≥ 2 (at Least Moderately Improved From Baseline) at Day 90
Description: The participants assessed the degree of change of their MMP using a single item composed of 7 grades (3 to -3) where: 3=much improved, 2=moderately improved, 1=minimally improved, 0=no change, -1=minimally worse, -2=moderately worse, and -3=much worse. The percentage of participants where the participant selected 2=moderately improved, or 3=much improved as compared to Baseline are reported.
Time Frame: Baseline (Day 1) to Day 90
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX® 48U | BOTOX® 72U
Number analyzed (Participants) | 46 | 53 | 46
percentage of participants | 21.7 [9.8 to 33.7] | 90.6 [82.7 to 98.4] | 73.9 [61.2 to 86.6]
Statistical Analysis 1: Comparison: Placebo vs BOTOX® 48U; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel — P-values for between-treatment comparisons are based on CMH model stratified by baseline MMPS Grade (4 or 5); Percentage Difference = 68.8, 95% CI 2-sided [54.5 to 83.1]
Statistical Analysis 2: Comparison: Placebo vs BOTOX® 72U; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel — P-values for between-treatment comparisons are based on CMH model stratified by baseline MMPS Grade (4 or 5); Percentage Difference = 52.2, 95% CI 2-sided [34.8 to 69.6]

11. Secondary Outcome: Change From Baseline in Lower Facial Volume at Day 90 Using Landmark Area of Interest (AOI) Analysis
Description: Lower facial volume was calculated from 3-dimensional (3D) surface images captured at Baseline and Day 90. The analysis region is defined using a series of anatomical landmarks placed on the baseline surface that are then projected mathematically to the posttreatment surface and verified by a technician. The difference in volume is measured between the select region of the baseline surface to the posttreatment surface. The lower facial volume is summed for both the left side and the right side of the face. An analysis of covariance (ANCOVA) model was used for analyses.
Time Frame: Baseline (Day 1) to Day 90
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: cubic centimeter (cm^3)
Arm/Group | Placebo | BOTOX® 48U | BOTOX® 72U
Number analyzed (Participants) | 46 | 53 | 46
cubic centimeter (cm^3) | -0.33 (0.511) | -6.15 (0.475) | -6.14 (0.505)
Statistical Analysis 1: Comparison: Placebo vs BOTOX® 48U; Test type: Superiority; p < .0001, ANCOVA — The change from baseline was analyzed using ANCOVA with study intervention and investigator site as factors and baseline MMPS Grade as a covariate; Least Squares (LS) Mean Difference = -5.82, 95% CI 2-sided [-7.10 to -4.54], Standard Error of Mean 0.647
Statistical Analysis 2: Comparison: Placebo vs BOTOX® 72U; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LS Mean Difference = -5.81, 95% CI 2-sided [-7.15 to -4.47], Standard Error of Mean 0.678

12. Secondary Outcome: Change From Baseline in Lower Facial Volume at Day 90 Using Statistical MMP AOI Analysis
Description: Lower facial volume was calculated from 3D surface models of the full area of the lower face captured at Baseline and Day 90. The statistical MMP AOI method is based on a statistical shape averaging of the area of change post masseter treatment from multiple facial models. The difference in volume is calculated between the two 3D surface models at Baseline and Day 90. An ANCOVA model was used for analyses.
Time Frame: Baseline (Day 1) to Day 90
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: cm^3
Arm/Group | Placebo | BOTOX® 48U | BOTOX® 72U
Number analyzed (Participants) | 46 | 53 | 46
cm^3 | -0.09 (0.598) | -7.72 (0.555) | -8.35 (0.590)
Statistical Analysis 1: Comparison: Placebo vs BOTOX® 48U; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LS Mean Difference = -7.63, 95% CI 2-sided [-9.12 to -6.13], Standard Error of Mean 0.756
Statistical Analysis 2: Comparison: Placebo vs BOTOX® 72U; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LS Mean Difference = -8.26, 95% CI 2-sided [-9.83 to -6.69], Standard Error of Mean 0.793

ADVERSE EVENTS:
Time Frame: First dose (Day 1) to the End of Study (Up to Day 180)
Arm/Group | Placebo | BOTOX® 48U | BOTOX® 72U
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/53 | 0/49
Serious Adverse Events (participants affected / at risk) | 1/48 | 1/53 | 0/49
Other Adverse Events (participants affected / at risk) | 0/48 | 6/53 | 4/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | BOTOX® 48U (N=53) | BOTOX® 72U (N=49)
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | BOTOX® 48U (N=53) | BOTOX® 72U (N=49)
Nasopharyngitis (Infections and infestations) | 0 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT03861936/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT03861936/SAP_001.pdf